CLINICAL TRIAL: NCT01279187
Title: The Impact of Parathyroid Hormone (PTH) on Craniofacial Osseous Regeneration in Bone
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was terminated due to patient complications unrelated to study drugs
Sponsor: University of Michigan (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Principal Investigator, Jill Bashutski, Clinical Assistant Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HUM00042770
Record Dates: First submitted 2011-01-18; First posted 2011-01-19 (Estimated); Results first posted 2018-02-07 (Actual); Last update posted 2018-02-07 (Actual); Status verified 2018-01

CONDITIONS: Implant
Keywords: dental; implant
MeSH Terms: interventions — Teriparatide; Carrier State

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Teriparatide (Experimental): demeclocycline HCl (150 mg, four times per day for 3d) followed by a 12 day intermission then 3 more days of demeclocycline HCl (150 mg, four times per day). One day after the last demeclocycline dosage, subjects will be instructed to self-administer teriparatide (or placebo) for 7 weeks. Twenty-five days after the last demeclocycline dosage, subjects will begin their second set of tetracycline labels:(250 mg, four times per day) for three days, followed by 12 days off, and then repeat another 3 days of tetracycline HCl (250 mg, four times per day). On day of the last teriparatide (or placebo) injection, subjects will present for bone core removal and dental implant placement.
  Interventions: Drug: Teriparatide
- Control (Placebo Comparator): demeclocycline HCl (150 mg, four times per day for 3d) followed by a 12 day intermission then 3 more days of demeclocycline HCl (150 mg, four times per day). One day after the last demeclocycline dosage, subjects will be instructed to self-administer teriparatide (or placebo) for 7 weeks. Twenty-five days after the last demeclocycline dosage, subjects will begin their second set of tetracycline labels:(250 mg, four times per day) for three days, followed by 12 days off, and then repeat another 3 days of tetracycline HCl (250 mg, four times per day). On day of the last teriparatide (or placebo) injection, subjects will present for bone core removal and dental implant placement.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Teriparatide — 20ug per day,via subcutaneous injection, for 7 weeks
  Other Names: Forteo
  Arms: Teriparatide
Drug: Placebo — 20ug per day, self administered injection, for 7 weeks
  Other Names: carrier
  Arms: Control

SUMMARY:
Good bone healing and bone build-up are necessary for the success of dental implants. Research in animals and humans has shown that a drug, called Forteo, can increase bone build-up and bone strength over time. Forteo has been approved by the Food and Drug Administration (FDA) for use in patients with a condition where bone is broken down and weakened, called osteoporosis. The investigators do not know, however, whether Forteo is effective for use in humans for improving bone healing after implant placement, and whether it will have the same bone-building and bone-strengthening effects as for patients with osteoporosis. This research study is being done to learn what effect 7 weeks of treatment with Forteo will have on bone build-up and strengthening of bone for patients receiving implants.

DETAILED DESCRIPTION:
A single center, placebo-controlled, double blind parallel study of teriparatide use in patients requiring dental implant therapy is planned. Subjects who qualify based on the inclusion/exclusion criteria will be randomly placed into one of two treatment groups, teriparatide (20 μg/day) or placebo control. Both patients and investigators will be blinded. Serum and gingival crevicular fluid (GCF) samples, radiographs, and a tetracycline-labelled bone core will constitute the main data gathered for analysis. After implant surgery, patients will return at 2 weeks for post-operative care and then at 14 weeks for an implant impression and again at 16 weeks to receive the final restoration. Twelve months after implant placement, patients will be seen for a follow-up exam and standardized radiograph to ensure proper healing.

ELIGIBILITY:
Inclusion Criteria:

* Age range 30-85 yrs
* Sex: male and female (female subjects must be postmenopausal, surgically sterilized or utilizing birth control or abstinence throughout the period of Teriparatide administration)
* Subjects must be able and willing to follow study procedures and instructions;
* Subjects must have read, understood and signed an informed consent form;
* Subjects must have a need for the replacement of at least one tooth in the mandibular premolar/molar region with at least 12 months since the tooth extraction.
* Sites must be adaptable for dental implant placement without the necessity for grafting.

Exclusion Criteria:

* Subjects under 30 years or over 85 years of age,
* Female subjects who are pregnant, lactating, or female subjects who are of childbearing potential who are not using contraceptives,
* Subjects with metabolic bone diseases such as Paget's disease, hypercalcemia (mild to moderate hypocalcemia is acceptable for entry into the study), moderate to severe vitamin D3 abnormalities (If vitamin D levels are below 16 ng/ml and patient exhibits interest, dietary supplementation will be suggested and levels re-evaluated after 4 weeks and reconsidered for inclusion at that time), any other metabolic bone diseases including osteoporosis,
* Subjects with prior radiation therapy, bone metastases or other skeletal malignancy,
* Subjects on medications that would affect bone metabolism,
* Subjects with growth hormone deficiency,
* Subjects with uncontrolled diabetes, sprue, inflammatory bowel disease or other disorders that would affect calcium absorption
* Subjects that are heavy smokers (> 1 pack/d),
* Subjects with tetracycline sensitivity or allergy,
* Subjects on bisphosphonates,
* Subjects with any form of kidney disease including kidney stones (urolithiasis and nephrolithiasis),
* Subjects with known allergies to tetracycline and/or demeclocycline,

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2011-02; Primary Completion 2015-03 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jill Bashutski, DDS, MS, Principal Investigator — Faculty
Locations (1):
- Michigan Center for Oral Health Research, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hanley, D., et al., Pharmacologic mechanisms of therapeutics:Parathyroid Hormone, in Principles of Bone Biology, J. Bilezikian, L. Raisz, and T. Martin, Editors. 2008, Academic Press: San Diego. p. 1661-1695.
- [Background] Neer RM, Arnaud CD, Zanchetta JR, Prince R, Gaich GA, Reginster JY, Hodsman AB, Eriksen EF, Ish-Shalom S, Genant HK, Wang O, Mitlak BH. Effect of parathyroid hormone (1-34) on fractures and bone mineral density in postmenopausal women with osteoporosis. N Engl J Med. 2001 May 10;344(19):1434-41. doi: 10.1056/NEJM200105103441904. PMID 11346808
- [Background] Alkhiary YM, Gerstenfeld LC, Krall E, Westmore M, Sato M, Mitlak BH, Einhorn TA. Enhancement of experimental fracture-healing by systemic administration of recombinant human parathyroid hormone (PTH 1-34). J Bone Joint Surg Am. 2005 Apr;87(4):731-41. doi: 10.2106/JBJS.D.02115. PMID 15805200
- [Background] Chen H, Frankenburg EP, Goldstein SA, McCauley LK. Combination of local and systemic parathyroid hormone enhances bone regeneration. Clin Orthop Relat Res. 2003 Nov;(416):291-302. doi: 10.1097/01.blo.0000079443.64912.18. PMID 14646773

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Teriparatide | Control
Started | 14 | 13
Completed | 14 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Teriparatide | Control | Total
Number analyzed (Participants) | 14 | 13 | 27
Age, Continuous [Mean (Full Range); unit: years] | 54 [33 to 71] | 53.5 [33 to 71] | 53.95 [33 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 6 | 15
  Male | 5 | 7 | 12
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 14 | 13 | 27

OUTCOME MEASURES:

1. Primary Outcome: Bone Formation Rate
Description: To determine the impact of PTH on bone quality and bone turnover in the oral cavity. The primary outcome variable will be bone formation rate.
Time Frame: 10 weeks
Measure: Median (Standard Deviation); unit: mm2/week
Arm/Group | Teriparatide | Control
Number analyzed (Participants) | 14 | 13
mm2/week | 1.76 (0.99) | 2.22 (1.67)

2. Secondary Outcome: Bone Turnover (Mineral Apposition Rates)
Description: Bone turnover was assessed indirectly by bone histomorphometry using the following abbreviations: Mineral Apposition Rate (MAR): Distance between 2 fluorochrome markers that comprise a double label on the surfaces of cancellous bone measured at an average of 4 equally-spaced sites per double label. These measurements will be performed on 20 double fluorochrome labels per bone and the average divided by the time between the midpoints of the two labeling periods. MAR serves as an index of osteoblast activity. Reported for cancellous (Cn), endocortical (Ec) at baseline (pre-drug intervention, listed as "first set") and at the end of drug intervention ("second set"). "First set" refers to baseline information (pre-drug), and "second set" refers to data evaluated at the end of the drug administration phase. Periosteal (Ps) data and Ec.Mar Endocortical MAR "second set" was reviewed but no analyzable labeling was noted and so this data is not reported.
Time Frame: 10 weeks
Measure: Mean (Standard Deviation); unit: um/day
Arm/Group | Teriparatide | Control
Number analyzed (Participants) | 14 | 13
um/day
  Cn.MAR (Cancellous MAR) - first set | 0.5 (0.1) | 0.3 (0.2)
  Ec.MAR Endocortical MAR - first set | 0.7 (0.7) | 0.6 (0.4)
  Cn.MAR Cancellous MAR- second set | 0.2 (0.2) | 0.3 (0.2)

3. Secondary Outcome: Bone Turnover: Cortical Tissue Area
Description: Bone turnover was assessed indirectly by evaluating cellular parameters of PTH action (i.e. numbers of osteoblasts, osteoclasts, apoptotic osteoblasts). The methods used to obtain the outcomes described below were bone histomorphometry using the following abbreviation:
  Ct.T.Ar: Ct Cort(ex)(ical) Tissue Area (2D)b "First set" refers to baseline pre-drug data and "second set" was taken at the end of the drug administration phase.
Time Frame: 10 weeks
Measure: Mean (Standard Deviation); unit: mm2/week
Arm/Group | Teriparatide | Control
Number analyzed (Participants) | 14 | 13
mm2/week
  Ct.T.Ar first set Cortical Tissue Area | 2.2 (1.6) | 1.8 (1)
  Ct. T.Ar second set Cortical Tissue Area | 2.2 (1.6) | 1.8 (0.9)

4. Secondary Outcome: Bone Turnover: Bone Perimeter Length
Description: Bone histomorphometry was used to assess bone perimeter length in mm as follows:
  Cn.Pm cancellous: Cancellous Bone Perimeter Ec.Pm: endocortical bone perimeter Ps.Pm: Periosteal Periosteal bone perimeter
Time Frame: 10 weeks
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Teriparatide | Control
Number analyzed (Participants) | 14 | 13
mm
  Cn.Pm cancellous Cancellous bone Perimeter | 20.8 (11.1) | 18.7 (9.6)
  Ec.Pm endocortical bone perimeter | 2.9 (1.5) | 3.6 (1.3)
  Ps.Pm Periosteal Periosteal bone perimeter | 4.1 (0.9) | 4.3 (1.1)

5. Secondary Outcome: Bone Turnover: Bone Percentages
Description: Oc.S/BS cancellous: Osteoclast suface divided by bone surface. Osteoclastic surface as percent of total bone surface in cancellous bone. Percent cancellous bone perimeter with osteoclasts (large, multinuclear, TRAP positive cells).
  OS/BS cancellous: Osteoid surface divided by bone surface. Percentage of cancellous bone perimeter covered with osteoid.
  Oc.S/BS endocortical: Osteoclastic surface as percent of total bone surface in endocortical bone.
  OS/BS endocortical: Percentage of endocortical bone perimeter covered with osteoid.
  Oc.S/BS Periosteal: Osteoclastic surface as percent of total bone surface in periosteal bone.
  Ob.S/BS Periosteal: Percent periosteal bone perimeter with osteoid and adjacent osteoblasts, identified as plump cells with a single, eccentric nucleus and a pale-staining golgi apparatus. Osteoblast Surface divided by bone surface in periosteal bone.
  OS/BS Periosteal: Percentage of periosteal bone perimeter covered with osteoid.
Time Frame: 10 weeks
Measure: Mean (Standard Deviation); unit: percentage (%)
Arm/Group | Teriparatide | Control
Number analyzed (Participants) | 14 | 13
percentage (%)
  Oc.S/BS cancellous | 0.34 (0.42) | 0.15 (0.21)
  OS/BS cancellous | 8 (10) | 12 (11)
  Oc.S/BS endocortical | 0 (0) | 0.3 (0.7)
  OS/BS endocortical | 14 (27) | 17 (23)
  Oc.S/BS Periosteal | 0.1 (0.2) | 0.4 (1.2)
  Ob.S/BS Periosteal | 6 (13) | 5 (11)
  OS/BS Periosteal | 5 (22) | 25 (28)

ADVERSE EVENTS:
Time Frame: 59 weeks
Arm/Group | Teriparatide | Control
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/13
Other Adverse Events (participants affected / at risk) | 12/14 | 11/13
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Teriparatide (N=14) | Control (N=13)
Debonded Crown (General disorders) | 3 (4) | 8 (13) — Implant crown came off
Implant Failure (General disorders) | 4 (4) | 6 (6)
Thrush (General disorders) | 1 (1) | 0 (0)
Shingles (General disorders) | 0 (0) | 1 (1)
Sore Throat (General disorders) | 1 (2) | 0 (0)
Metallic taste (General disorders) | 0 (0) | 1 (1)
Leg Cramps (General disorders) | 1 (1) | 0 (0)
Constipation (General disorders) | 0 (0) | 1 (1)
Joint pain (General disorders) | 0 (0) | 2 (2)
Indigestion (General disorders) | 1 (2) | 0 (0)
Discontinuation of Drug (General disorders) | 0 (0) | 1 (1) — Patient chose to stop taking the drug without informing the study team
Flu (General disorders) | 1 (1) | 1 (1)
headache (General disorders) | 1 (1) | 0 (0)
rotator cuff injury (General disorders) | 1 (1) | 0 (0)
Pt received tetanus shot (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No